CLINICAL TRIAL: NCT06456047
Title: Detection of Early Airway Obstruction in Patients with Chronic Obstructive Pulmonary Disease Using Expiratory Time Constant
Brief Title: Detection of Early Airway Obstruction in Patients with COPD Using RCexp
Acronym: COPD TiCON
Status: Not yet recruiting | Type: Observational
Sponsor: East Slovak Institute for Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Filip Depta MD, MD, PhD, East Slovak Institute for Cardiovascular Diseases
Other Study IDs: VUSCH
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; expiratory time constant
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all patients undergoing routine spirometry: all patients undergoing routine spirometry and have GOLD or STAR negative criteria but positive RCexp

SUMMARY:
We hypothesize that Cexp during tidal and forced exhalation implemented to the routine spirometer may detect airway obstruction earlier than conventional spirometric indices such as FEV1 and FEV1/FVC.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the most common chronic lung disease worldwide, leading to significant morbidity, mortality, and high treatment costs. In 2020, the global prevalence of COPD was estimated to be 10.6%, affecting around 480 million people. The diagnosis of COPD in suspected patients is typically confirmed through routine spirometry, a simple noninvasive test that assesses the degree of airway obstruction. However, research has revealed that extensive small airway disease exists in COPD before it can be detected using traditional spirometric measures, such as forced expiratory volume in the first second (FEV1) and the ratio of FEV1 to forced expiratory capacity (FEV1/FVC). Efforts are underway to find new parameters to improve early detection of airway obstruction in patients with COPD. The expiratory time constant (RCexp) is a promising variable studied in critical care medicine and may also prove useful in pulmonology. Data from ventilated COPD patients demonstrate that prolonged RCexp was present in all patients with COPD. The FEV1/FVC ratio is currently the gold standard for diagnosing COPD, but it only yields a single calculated value. In contrast, RCexp may offer more precision as it reflects exhalation dynamics at multiple time points during exhalation. If there is a prolongation of subsequent RCexp towards the end of exhalation, it could indicate the presence of obstruction. We hypothesize that RCexp during tidal and forced exhalation implemented to the routine spirometer may detect airway obstruction earlier than conventional spirometric indices such as FEV1 and FEV1/FVC.

ELIGIBILITY:
Inclusion Criteria: all patients eligible for routine spirometry if indicated as per the standard of care -

Exclusion Criteria: known pulmonary disease, post thoracic surgery

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients that are subjected to routine spirometry
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of early airway obstruction and positivity of RCexp | January 2025 - December 2028
  research correlation of RCexp1, RCexp2, and RCexp3 with FEV1 and FEV1/FVC in patients with known COPD and its correlation with healthy controls

IPD SHARING:
Plan to Share IPD: Undecided
Depending on secondary data analyses

REFERENCES:
- [Background] Depta F, Euliano NR, Zdravkovic M, Torok P, Gentile MA. Time constant to determine PEEP levels in mechanically ventilated COVID-19 ARDS: a feasibility study. BMC Anesthesiol. 2022 Dec 13;22(1):387. doi: 10.1186/s12871-022-01935-8. PMID 36513978